CLINICAL TRIAL: NCT04042103
Title: Open-Label Maximal Use Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Tapinarof Cream, 1% in Adults With Extensive Plaque Psoriasis
Brief Title: Maximal Use Study of Tapinarof Cream, 1% in Adults With Extensive Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMVT-505-2002
Record Dates: First submitted 2019-07-24; First posted 2019-08-01 (Actual); Results first posted 2022-05-06 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2022-05

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: Open-label, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tapinarof (DMVT-505) cream, 1% (Experimental): Tapinarof (DMVT-505) cream, 1% applied topically once daily
  Interventions: Drug: Tapinarof cream, 1%

INTERVENTIONS:
Drug: Tapinarof cream, 1% — Tapinarof cream, 1% applied topically once daily
  Other Names: DMVT-505

SUMMARY:
This is an open-label, multicenter study to evaluate the systemic exposure and safety of topical tapinarof cream, 1% under conditions of maximal use in adults with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 18 to 75 with a confirmed clinical diagnosis of plaque psoriasis and stable disease for at least 6 months prior to the study
* BSA involvement ≥ 20%
* PGA score of ≥ 3 at screening
* Females of child bearing potential and male subjects who are engaging in sexual activity that could lead to pregnancy agree to follow the specified contraceptive guidance throughout the study
* Capable of giving written informed consent

Exclusion Criteria:

* Psoriasis other than plaque variant
* Any sign of infection of any of the psoriatic lesions
* Evidence of significant hepatic, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular (CV) system abnormalities or laboratory abnormality that will affect the health of the subject or interfere with the interpretation of the results
* Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation within 4 weeks prior to the Baseline visit and/or plans to have such exposures during the study which could potentially impact the subject's psoriasis
* Use of any prohibited medication within the indicated period before the first dose of study drug
* Pregnant females or lactating females
* The subject has received an investigational product within 30 days, 5 half-lives, or twice the duration of the biological effect of the study drug (whichever is longer) prior to first dose of study drug
* Current or a history of cancer within 5 years except for fully excised skin basal cell carcinoma, squamous cell carcinoma or carcinoma in situ of the cervix
* Previous known participation in a clinical study with tapinarof

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael McLaughlin, Study Director — Dermavant Sciences, Inc.
Locations (6):
- United States (6):
  - Dermavant Investigational Site, Encino, California
  - Dermavant Investigational Site, Sanford, Florida
  - Dermavant Investigational Site, Philadelphia, Pennsylvania
  - Dermavant Investigational Site, Austin, Texas
  - Dermavant Investigational Site, San Antonio, Texas
  - Dermavant Investigational Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jett JE, McLaughlin M, Lee MS, Parish LC, DuBois J, Raoof TJ, Tabolt G, Wilson T, Somerville MC, DellaMaestra W, Piscitelli SC. Tapinarof Cream 1% for Extensive Plaque Psoriasis: A Maximal Use Trial on Safety, Tolerability, and Pharmacokinetics. Am J Clin Dermatol. 2022 Jan;23(1):83-91. doi: 10.1007/s40257-021-00641-4. Epub 2021 Oct 28. PMID 34713415

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Started | 21
Completed | 19
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Adverse Events (AEs), Severe Adverse Events, and Serious Adverse Events (SAEs)
Description: Frequency and severity of AEs (local and systemic)
Time Frame: Baseline to Week 4
Population: Safety Analysis Set: All randomized subjects who receive at least 1 application of study drug will be included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
Participants
  Experienced an AE | 12
  Experienced a Treatment-Related AE | 6
  Experienced a Grade 3 (severe) AE | 2
  Experienced a Grade 4 (life-threatening) AE | 0
  Experienced a Grade 5 (fatal) AE | 0
  Experienced an SAE | 1
  Experienced a Treatment-related SAE | 0
  Experienced TEAE leading to discontinuation from study/drug | 0

2. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Values, Biomarker Values, ECG Results or Vital Signs
Description: Changes in laboratory values, biomarker values, ECG results and vital signs were assessed for clinical relevance.
Time Frame: Baseline to Week 4 or Follow-Up (7-10 days after Week 4 Visit)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
Participants
  Clinically Meaningful changes in hematology. | 0
  Clinically meaningful changes in chemistry | 0
  Clinically meaningful changes in urinalysis | 0
  Clinically meaningful changes in tryptase | 0
  Clinically meaningful changes in ECG parameters | 0
  Clinically meaningful changes in vital signs | 0

3. Primary Outcome: Number of Participants With Irritation as Assessed by the Local Tolerability Scale
Description: At each specified study visit, the Investigator (or qualified evaluator) assessed the presence and overall degree of irritation at the application sites, according to the LTS. The score will ideally represent an 'average' across all application sites. To the fullest extent possible, the same Investigator (or designated evaluator) will perform all tolerability assessments for an individual participant throughout the study.
Time Frame: Day 1, Day 15, Day 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
Participants
  Baseline: No Irritation | 14
  Baseline: Mild | 5
  Baseline: Moderate | 1
  Baseline: Severe | 1
  Baseline: Very Severe | 0
  Day 15: number analyzed (Participants) | 20
  Day 15: No Irritation | 14
  Day 15: Mild | 5
  Day 15: Moderate | 1
  Day 15: Severe | 0
  Day 15: Very Severe | 0
  Day 29: number analyzed (Participants) | 19
  Day 29: No Irritation | 17
  Day 29: Mild | 2
  Day 29: Moderate | 0
  Day 29: Severe | 0
  Day 29: Very Severe | 0

4. Primary Outcome: Tapinarof and Tapinarof Sulfate (Metabolite) Plasma PK Parameters on Day 1 and Day 29: AUCo-tau
Description: The AUC in plasma is a pharmacokinetic parameter that describes the overall exposure of the drug.
Time Frame: Day 1 and Day 29 (PK samples collected at pre-dose and at 1, 2, 3, 4, 5, 8, 12, and 24 hours after dosing)
Population: PK Analysis set: All subjects who have at least 1 application of study drug and have at least 1 evaluable PK assay result will be included in the PK analysis set. The majority of subjects had plasma levels of tapinarof and tapinarof sulfate that were below the level of quantitation (BQL). AUCo-tau value could not be calculated for 17 of the 21 subjects on Day 1 and 18 of the 19 subjects on Day 29, due to BQL samples. The metabolite (tapinarof sulfate) was BQL in all samples.
Measure: Mean (Standard Error); unit: pg*h/ml
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
pg*h/ml
  Day 1: tapinarof: number analyzed (Participants) | 4
  Day 1: tapinarof | 8037.29 (6204.935)
  Day 29: tapinarof: number analyzed (Participants) | 1
  Day 29: tapinarof | 1985.54 (NA) — Subjects with a minimum of 3 postdose time points were required for determination of AUC. N=1 for Day 29

5. Primary Outcome: Tapinarof and Tapinarof Sulfate (Metabolite) Plasma PK Parameters on Day 1 and Day 29: Cmax
Description: The Cmax is a pharmacokinetic parameter that describes the highest concentration of the drug that is achieved after dosing.
Time Frame: Day 1 and Day 29 (PK samples collected at pre-dose and at 1, 2, 3, 4, 5, 8, 12, and 24 hours after dosing)
Population: PK Analysis Set: All subjects who have at least 1 application of study drug and have at least 1 evaluable PK assay result will be included in the PK analysis set. No subject had measurable concentrations of the metabolite (tapinarof sulfate) at any time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
pg/mL
  Day 1: tapinarof Cmax | 898.33 (1448.084)
  Day 29: tapinarof Cmax: number analyzed (Participants) | 19
  Day 29: tapinarof Cmax | 116.09 (148.424)

6. Primary Outcome: Tapinarof and Tapinarof Sulfate (Metabolite) Plasma PK Parameters on Day 1 and Day 29: Tmax and t1/2
Description: The tmax is a pharmacokinetic parameter that describes the time point at which the highest concentration of the drug is achieved after dosing.
Time Frame: Day 1 and Day 29 (PK samples collected at pre-dose and at 1, 2, 3, 4, 5, 8, 12, and 24 hours after dosing)
Population: PK Analysis Set: All subjects who have at least 1 application of study drug and have at least 1 evaluable PK assay result were included in the PK analysis set. No subject had measurable concentrations of the metabolite (tapinarof sulfate) at any time point. An elimination half-life (t½) could not be determined in the majority of subjects (19/21 subjects [90.5%]) on Day 1 and all subjects on Day 29 due to the lack of detectable tapinarof in plasma samples in the elimination phase.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
hours
  Day 1: tmax: number analyzed (Participants) | 18
  Day 1: tmax | 4.39 (5.476)
  Day 29: tmax: number analyzed (Participants) | 11
  Day 29: tmax | 4.02 (3.005)
  Day 1: t1/2: number analyzed (Participants) | 2
  Day 1: t1/2 | 6.41 (0.691)

7. Secondary Outcome: Change From Baseline in QTcF (ΔQTcF) at Each Post-treatment Time Point on the Sampling Day With the Higher Cmax (Day 1 or Day 29)
Description: Identify clinically relevant effect of tapinarof on cardiac conduction
Time Frame: Baseline and Day 1
Population: QT/QTc analysis set: The QT/QTc analysis set will include all subjects in the safety analysis set with measurements at Baseline as well as on-treatment with at least 1 post-dose time point with a valid ΔQTcF value.
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
ms
  Day 1 1 h Post-dose: number analyzed (Participants) | 20
  Day 1 1 h Post-dose | -7.2 (1.79)
  Day 1 2 h Post-dose | -1.1 (2.92)
  Day 1 3 h Post-dose: number analyzed (Participants) | 19
  Day 1 3 h Post-dose | -4.3 (1.88)
  Day 1 4 h Post-dose: number analyzed (Participants) | 20
  Day 1 4 h Post-dose | -2.3 (3.04)
  Day 1 5 h Post-dose: number analyzed (Participants) | 18
  Day 1 5 h Post-dose | -4.9 (2.87)
  Day 1 8 h Post-dose: number analyzed (Participants) | 20
  Day 1 8 h Post-dose | -3.0 (2.60)
  Day 1 12 h Post-dose: number analyzed (Participants) | 19
  Day 1 12 h Post-dose | -1.6 (2.18)
  Day 1 24 h Post-dose | -3.4 (1.97)

8. Secondary Outcome: Analysis of the Relationship Between Plasma Concentration and ΔQTcF
Description: The relationship between tapinarof plasma concentrations and ∆QTcF was investigated using a linear mixed-effects modeling approach with ΔQTcF as the dependent variable. A linear model with an intercept was fitted for tapinarof plasma concentrations, which represented the data in an acceptable way. The slope of tapinarof plasma concentration in the concentration-QTc relationship was estimated.
Time Frame: Day 1
Population: PK/QTc Analysis Set included all subjects with at least 1 pair of post-dose PK and QTcF data from the same time point.
  Of the 21 total subjects, there were 10, 8, 12, 10, 11, 11, 13, and 17 subjects with tapinarof plasma concentrations BLQ at the 1, 2, 3, 4, 5, 8, 12, and 24 hour post-dose time points, respectively. The number of participants with measurable tapinarof ranged from 4 to 13 across all the timepoints. The slope is determined based on the data available for each timepoint.
Measure: Number (90% Confidence Interval); unit: ms per pg/ml
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
ms per pg/ml | -0.00016 [-0.002172 to 0.001844]

9. Secondary Outcome: Mean Change From Baseline to Day 29 in Physician's Global Assessment (PGA)
Description: The PGA is a clinical tool for assessing the current state/severity of a subject's psoriasis at a given timepoint. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, scaling, and plaque thickness/elevation as guidelines. Higher PGA scores represent more severe disease. This scale ranges from 0 to 5, with 0 = best outcome.
Time Frame: Baseline to Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
score on a scale | -1.2 (1.03)

10. Secondary Outcome: Mean Change From Baseline to Day 29 Psoriasis Area and Severity Index (PASI)
Description: The Psoriasis Area and Severity Index (PASI) scoring system combines the assessment of lesion severity and extent of affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, and legs). Each area is assessed for 3 signs: erythema (redness), induration (plaque thickness), and scale. The severity of each sign in each body area is assessed and scored independently using a 5-point scale, where 0=none, 1=slight, 2=mild, 3=moderate, 4=severe. Each area is also assessed for percent of skin involved: 0 = (0%), 1 = (1-<10%), 2 = (10-<30%), 3 = (30-<50%), 4 = (50 -<70%), 5 = (70-<90%), 6 = (90-100%). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Time Frame: Baseline to Day 29
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
score on a scale | -15.14 [-19.61 to -10.66]

11. Secondary Outcome: Mean Change From Baseline to Day 29 in Percent of Total Body Surface Area (%BSA) Affected
Description: The assessment of %BSA affected is an estimate of the percentage of total involved skin with psoriasis. For the purpose of clinical estimation, the total palmar surface of the subject's palm and digits may be assumed to be approximately equivalent to 1% BSA. The %BSA affected by psoriasis will be evaluated (from 0% to 100%). %BSA is a static assessment made without reference to previous scores.
Time Frame: Baseline to Day 29
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of BSA affected
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
Number analyzed (Participants) | 21
percentage of BSA affected | -14.44 [-19.84 to -9.04]

ADVERSE EVENTS:
Time Frame: Study Period (29 days) + Follow-up period (7 to 10 days)
Arm/Group | Tapinarof (DMVT-505) Cream, 1%
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 12/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapinarof (DMVT-505) Cream, 1% (N=21)
pancreatitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapinarof (DMVT-505) Cream, 1% (N=21)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Folliculitis (Infections and infestations) | 4 (4)
Furuncle (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT04042103/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT04042103/SAP_001.pdf